CLINICAL TRIAL: NCT00573222
Title: Non-interventional Surveillance of Effectiveness of Symbicort® Maintenance And Reliever Therapy (Symbicort® SMART) in the Treatment of Moderate and Severe Asthma
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-RHR-SYM-2007/1
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Symbicort

SUMMARY:
This is a 3-month non-interventional, observational study on patients with moderate and severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate and severe asthma on Symbicort SMART treatment

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pulmonology clinics
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To evaluate & describe asthma control in adult patients w/moderate to severe asthma treated w/Symbicort SMART following the frequency, type & severity of symptoms through the Asthma Control Questionnaire.

SECONDARY OUTCOMES:
to evaluate the safety of Symbicort SMART treatment through the number and type of reported adverse events 2. assessment of patient's satisfaction with the treatment 3.assessment of physician's satisfaction with the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anan Marija Gjurovic, Study Director — AstraZeneca
Locations (13):
- Croatia (13):
  - Research Site, Čakovec
  - Research Site, Dubrovnik
  - Research Site, Osijek
  - Research Site, Požega
  - Research Site, Pula
  - Research Site, Rijeka
  - Research Site, Senj
  - Research Site, Slavonskibrod
  - Research Site, Šibenik
  - Research Site, Vinkovci
  - Research Site, Vukovar
  - Croatia, Zadar
  - Research Site, Zagreb